CLINICAL TRIAL: NCT05409404
Title: The Effects of 8 Weeks Post Exercise Hot Water Immersion on Vascular and Cardiometabolic Health in Physically Inactive Middle-aged Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coventry University (Other)
Collaborators: British Society for Research on Ageing (Unknown)
Responsible Party: Principal Investigator, Charles Steward, Post Graduate Research Student, Coventry University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P132234
Record Dates: First submitted 2022-03-18; First posted 2022-06-08 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Physical Inactivity; Aging
MeSH Terms: conditions — Sedentary Behavior | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic exercise + hot water immersion (Experimental): 3 sessions per week, over an 8 week period, with each session consisting of 30 minutes of aerobic exercise (10 minutes cycling, jogging and rowing) at a power output equivalent to 65-75% of maximal heart rate followed by 30 minutes of whole body hot water immersion at 40°C.
  Interventions: Other: Aerobic exercise + hot water immersion
- Aerobic exercise + thermoneutral water immersion (Active Comparator): 3 sessions per week, over an 8 week period, with each session consisting of 30 minutes of aerobic exercise (10 minutes cycling, jogging and rowing) at a power output equivalent to 65-75% of maximal heart rate followed by 30 minutes of whole body water immersion at 34°C.
  Interventions: Other: Aerobic exercise + thermoneutral water immersion

INTERVENTIONS:
Other: Aerobic exercise + hot water immersion — Light to moderate intensity aerobic exercise for 30 minutes, followed by 30 minutes of hot water immersion at 40°C.
  Arms: Aerobic exercise + hot water immersion
Other: Aerobic exercise + thermoneutral water immersion — Light to moderate intensity aerobic exercise for 30 minutes, followed by 30 minutes of thermoneutral water immersion at 34°C.
  Arms: Aerobic exercise + thermoneutral water immersion

SUMMARY:
This research project aims to determine whether post exercise hot water immersion can improve vascular and cardiometabolic health to a greater extent than post exercise thermoneutral water immersion in healthy middle-aged adults.

The study will take place over an 8 week period where participants will do a combination of aerobic exercise and water immersion 3 times per week. The study will be a randomised controlled trial comparing 8-weeks of post exercise hot water immersion (EX+HWI) to post exercise thermoneutral water immersion (EX+TNWI).

DETAILED DESCRIPTION:
The exercise component of each intervention will be 30 minutes of moderate intensity aerobic exercise consisting of 10 minutes cycling, jogging and rowing, three times per week. Exercise intensity will be maintained at a heart rate equivalent of 65% of maximal heart rate. All exercise sessions will take the form of supervised group exercise sessions (<4 participants) at Coventry University. After 30 minutes of exercise, participants will either complete 30 minutes of whole-body hot water immersion at 40°C or thermoneutral immersion at 34°C in the control condition (similar protocols are known to be well tolerated in older adults) (Akerman et al. 2019; Brunt et al. 2016). In order to ensure progression, exercise intensity will be increase to 75% of maximal heart rate according to the maximal exercise test at 4 weeks.

Assessment sessions will take place before session 1 and >48hrs after session 12 and 24. Prior to arriving at the lab participants will complete an overnight fast. Participants will also refrain from consuming alcoholic and caffeinated beverages, nitrate high sources and any form of strenuous exercise in the 24hr time period prior to testing. All testing laboratory visits will be completed in the morning and where possible at the same time of day to help standardise for any potential variations that the circadian rhythm may have on the measured variables.

Assessments will be completed over two days. The outcome measures for this study comprise a range of physiological psychological measures which are known to inform the risk of cardiovascular disease. These measures fall into the following broad categories 1) vascular health; 2) cardiometabolic and inflammatory blood markers; 3) maximal exercise test and 4) cardiovascular disease risk prediction. In addition, measures of intervention acceptability and basic physiological heat acclimation measures will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 45 - 65 years
* If female and post-menopausal (12 months without a period and not taking HRT)
* Body mass index (BMI) 18.5 - 34.9kg/m2
* Participated in less than 150 mins of moderate intensity physical activity or 75 mins of vigorous or a combination of both over the last 6 months.

Exclusion Criteria:

* Previous myocardial infarction or cerebrovascular event
* Any signs or symptoms of cardiovascular issues
* High blood pressure: SBP >180 mmHg and / or DBP >100 mmHg
* Orthostatic hypotension: Drop of SBP > 20mmHg and / or DBP >10 mmHg upon standing.
* Changed blood pressure medication in the 6-month period prior to the study
* Plan to change any form of relevant medication during study period
* Suffers from diabetes
* Suffers from severe asthma
* Currently have any infections or symptoms of an infection (e.g. COVID-19 etc)
* Suffers from a neurodegenerative disease
* Cannot understand and/or fully cooperate with the study protocol
* Exercise-limiting comorbidity (e.g. angina, chronic lung disease, arthritis etc)
* Severe peripheral neuropathy (cannot sense temperature)
* Current smoker or have stopped in the last 3 months
* Any skin conditions including ulcerations
* Exposed to high temperatures in the last 4-weeks (e.g. holiday, spa, sun beds etc)
* Use of antioxidant supplements in the last 6-weeks

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-01-13 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2023-08-25 (Actual)

PRIMARY OUTCOMES:
Change in resting systolic blood pressure (mmHg) | Measurements taken the week before the study, >48hrs after 4 weeks and >48hrs after 8 weeks
  Measured using an automated blood pressure cuff
Change in resting diastolic blood pressure (mmHg) | Measurements taken the week before the study, >48hrs after 4 weeks and >48hrs after 8 weeks
  Measured using an automated blood pressure cuff
Change in resting mean arterial blood pressure (mmHg) | Measurements taken the week before the study, >48hrs after 4 weeks and >48hrs after 8 weeks
  Measured using an automated blood pressure cuff
Change in flow mediated dilation (%) | Measurements taken the week before the study, >48hrs after 4 weeks and >48hrs after 8 weeks
  Terason ultrasound recording after brachial artery occlusion
Change in pulse wave velocity (ms-1) | Measurements taken the week before the study, >48hrs after 4 weeks and >48hrs after 8 weeks
  SphygmoCor XCEL measuring carotid to femoral arterial stiffness
Change in intima-media thickness (mm) | Measurements taken the week before the study, >48hrs after 4 weeks and >48hrs after 8 weeks
  Terason ultrasound image to measure wall thickness from the lumen-intima interface to the media-adventitia interface of the brachial and femoral arteries
Change in beta stifnness index | Measurements taken the week before the study, >48hrs after 4 weeks and >48hrs after 8 weeks
  Calculated using systolic, diastolic blood pressure from automated blood pressure cuff and vessel diameter from Terason ultrasound image of brachial and femoral arteries
Change in dynamic arterial compliance (mm2) | Measurements taken the week before the study, >48hrs after 4 weeks and >48hrs after 8 weeks
  Calculated using pulse pressure from automated blood pressure cuff and vessel diameter from Terasol ultrasound image of brachial and femoral arteries
Change in maximal oxygen uptake (ml/kg/min) | Measurements taken the week before the study, >48hrs after 4 weeks and >48hrs after 8 weeks
  Maximal oxygen uptake
Change in glucose tolerance (mmol/L) | Measurements taken the week before the study, >48hrs after 4 weeks and >48hrs after 8 weeks
  Oral glucose tolerance test through fingertip capillary blood samples at 15 minute intervals for the first 1 hour and 30 minute intervals for the second hour
Change in circulating serum Interleukin-6 (pg/ml) | Measurements taken the week before the study, >48hrs after 4 weeks and >48hrs after 8 weeks
  Venous blood sample
Change in circulating serum TNF-α (pg/ml) | Measurements taken the week before the study, >48hrs after 4 weeks and >48hrs after 8 weeks
  Venous blood sample
Change in circulating serum Interleukin-8 (pg/ml) | Measurements taken the week before the study, >48hrs after 4 weeks and >48hrs after 8 weeks
  Venous blood sample
Change in circulating serum Interleukin-10 (pg/ml) | Measurements taken the week before the study, >48hrs after 4 weeks and >48hrs after 8 weeks
  Venous blood sample
Change in circulating serum Interleukin-1Ra (pg/ml) | Measurements taken the week before the study, >48hrs after 4 weeks and >48hrs after 8 weeks
  Venous blood sample
Change in circulating Endothelin-1 (pg/ml) | Measurements taken the week before the study, >48hrs after 4 weeks and >48hrs after 8 weeks
  Venous blood sample
Circulating serum Monocyte chemoattractant protein-1 (pg/ml) | Measurements taken the week before the study, >48hrs after 4 weeks and >48hrs after 8 weeks
  Venous blood sample
Change in circulating serum Matrix metallopeptidase-2 (pg/ml) | Measurements taken the week before the study, >48hrs after 4 weeks and >48hrs after 8 weeks
  Venous blood sample
Change in circulating serum Matrix metallopeptidase-9 (pg/ml) | Measurements taken the week before the study, >48hrs after 4 weeks and >48hrs after 8 weeks
  Venous blood sample
Change in circulating total cholesterol (mmol/L) | Measurements taken the week before the study, >48hrs after 4 weeks and >48hrs after 8 weeks
  Venous blood sample
Change in circulating low density lipoproteins (mmol/L) | Measurements taken the week before the study, >48hrs after 4 weeks and >48hrs after 8 weeks
  Venous blood sample
Change in circulating high density lipoproteins (mmol/L) | Measurements taken the week before the study, >48hrs after 4 weeks and >48hrs after 8 weeks
  Venous blood sample
Change in circulating Triglycerides (mmol/L) | Measurements taken the week before the study, >48hrs after 4 weeks and >48hrs after 8 weeks
  Venous blood sample
Change in circulating glycated haemoglobin (%) | Measurements taken the week before the study, >48hrs after 4 weeks and >48hrs after 8 weeks
  Venous blood sample
Change in circulating basal glucose (mmol/L) | Measurements taken the week before the study, >48hrs after 4 weeks and >48hrs after 8 weeks
  Venous blood sample

SECONDARY OUTCOMES:
Change in Framingham risk score | Measurements taken the week before the study, >48hrs after 4 weeks and >48hrs after 8 weeks
  Calculation based on age, gender, total cholesterol, HDL cholesterol, smoker, diabetes status and systolic blood pressure
Change in rectal core temperature (°C) | Measurements taken the week before the study, >48hrs after 4 weeks and >48hrs after 8 weeks
  Measured using a rectal probe attached to a squirrel data logger
Change in resting heart rate (bpm) | Measurements taken the week before the study, >48hrs after 4 weeks and >48hrs after 8 weeks
  Measured using a heart rate monitor
Body mass index (kg/m²) | Measurements taken the week before the study, >48hrs after 4 weeks and >48hrs after 8 weeks
  Calculated through height and weight
Change in thermal comfort | Measurements taken pre and post visit 1, 12 (4 weeks) and 24 (8 weeks)
  Thermal comfort Likert scale from a positive score of +5 very comfortable (maximum) to a negative score of -5 very uncomfortable (minimum)
Change in thermal sensation | Measurements taken pre and post visit 1, 12 (4 weeks) and 24 (8 weeks)
  Thermal sensation Likert scale from a positive score of +5 hot (maximum) to a negative score of -5 cold (minimum)
Change in basic affect | Measurements taken pre and post visit 1, 12 (4 weeks) and 24 (8 weeks)
  Basic affect Likert scale from a positive score of +5 very good (maximum) to a negative score of -5 very bad (minimum)
Change in physical activity enjoyment | Measurements taken pre and post visit 1, 12 (4 weeks) and 24 (8 weeks)
  Feelings about exercise and / or passive heating on a Likert scale from a positive score of 1 (maximum) to a negative score of 7 (minimum)

CONTACTS AND LOCATIONS:
Locations (1):
- Coventry University, Coventry, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers. Data will be used to publish research articles in academic journals with all data fully anonymised.